CLINICAL TRIAL: NCT02409004
Title: A Phase I Study Assessing the Effects of Rifampin on the Pharmacokinetics of Ataluren in Healthy Subjects
Brief Title: Effects of Rifampin on the Pharmacokinetics of Ataluren
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-026-HV
Record Dates: First submitted 2015-03-24; First posted 2015-04-06 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: Drug-drug interaction
MeSH Terms: interventions — ataluren; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ataluren (Experimental): Ataluren 1375 mg powder for oral suspension administered once daily on Days 1 and 11 Rifampin 300 mg capsules administered twice daily on Day 3 to Day 12
  Interventions: Drug: Ataluren; Drug: Rifampin

INTERVENTIONS:
Drug: Ataluren — Powder for oral suspension (supplied in sachets) 1X 125 mg + 1 x 250 mg + 1000 mg (total of 1375 mg)
  Other Names: Ataluren(PTC124)
Drug: Rifampin — Capsule 2x3oo mg Oral
  Other Names: Rifadin®

SUMMARY:
This will be a single centre, Phase I, open-label, one cohort, one dose level, fixed-sequence, drug interaction study in healthy volunteers. The objective of this study is to determine the effects of rifampin on the pharmacokinetics of ataluren under fasting conditions.

DETAILED DESCRIPTION:
A total of 15 healthy, adult, male non-smokers, were included in this study. Subjects were administered ataluren on Day 1 followed by rifampin from Days 3 to12, and again ataluren on Day 11. On Day 11, ataluren was administered before rifampin administration.

Prior to entering the trial, subjects had a screening visit to establish eligibility within 28 days before study drug administration. Subjects were confined from at least10 hours before the first ataluren dosing on Day 1 until approximately 50 hours postdose(Day 3). Thereafter, subjects came back every morning from Days 4 to 10 for rifampin dosing. Then, subjects reported to the clinical site at least 10 hours before ataluren dosing on Day 11 (evening of Day 10) and remained in the clinical site until after 50 hours post-Day 11 ataluren dose (Day 13).

ELIGIBILITY:
Inclusion Criteria:

1. Male, non-smoker (no use of tobacco products within two years prior to screening), ≥18 and ≤55 years of age, with Body Mass Index (BMI) >20.0 and <30.0 kg/m2 and body weight ≥50.0 kg.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within four weeks prior to dosing. Subjects vomiting within 24 hours pre-first dose of ataluren will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the QI;
   2. the absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease;
   3. the absence of any known nonsense mutation-mediated disease including Duchenne Muscular Dystrophy.
3. Capable of consent.
4. Willing to take off dentures at dosing.
5. Consent to perform genotyping for UGT1A9

Exclusion Criteria:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen or urine cotinine test at screening.
3. History of allergic reactions to ataluren, rifampin, or other related drugs.
4. Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to the first study drug administration.
5. Any reason which, in the opinion of the QI, would prevent the subject from participating in the study.
6. Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
7. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
8. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within three months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], and crack) within one year prior to screening.
9. Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days (90 days for biologics) prior to the first dosing or concomitant participation in an investigational study involving no drug administration.
10. Use of medication other than topical products without significant systemic absorption:

    1. prescription medication within 14 days prior to the first dosing;
    2. over-the-counter products including natural health products (eg, food supplements and herbal supplements) within seven days prior to the first ataluren dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
    3. a depot injection or an implant of any drug within three months prior to the first dosing.
11. Donation of plasma within seven days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
12. Hemoglobin <128 g/L and hematocrit <0.37 L/L at screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 12 days
  The objective of this study is to determine the effects of rifampin on the pharmacokinetics of ataluren under fasting conditions.
Maximum plasma concentration (Cmax) | 12 days
  The objective of this study is to determine the effects of rifampin on the pharmacokinetics of ataluren under fasting conditions.

SECONDARY OUTCOMES:
Safety as measured by adverse events, laboratory abnormalities, vital signs, and electrocardiogram parameters | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Laskin, MD, Study Director — PTC Therapeutics
Locations (1):
- Inventiv, Québec, Canada

IPD SHARING:
Plan to Share IPD: No